CLINICAL TRIAL: NCT02845882
Title: Modified BFM (Berlin-Frankfurt-Munster)Backbone Therapy for Chinese Children or Adolescents With Newly Diagnosed Lymphoblastic Lymphoma
Brief Title: LBL-2016 for Children or Adolescents in China
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer Group, China (Network)
Collaborators: Shanghai Children's Medical Center (Other); Tongji Hospital (Other); West China Second University Hospital (Other); Qilu Hospital of Shandong University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Children's Hospital of Soochow University (Other); Nanjing Children's Hospital (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCG-LBL-2016
Record Dates: First submitted 2016-07-24; First posted 2016-07-27 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Prednisone; Vincristine; pegaspargase; Cytarabine; Cyclophosphamide; Daunorubicin; Mercaptopurine; Methotrexate; Dexamethasone; Doxorubicin; Vindesine; Ifosfamide; Etoposide; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low risk group (Other): Stage I or II: Induction I followed by extracompartmental Protocol M, and maintenance therapy for up to a total therapy duration of 96 weeks. Twenty triple intrathecal injections.
  Interventions: Drug: Prednisone,Vincristine, Pegylated-asparaginase, Cytarabine, Cyclophosphamide, Daunorubicin, 6-mercaptopurine; Drug: 6-mercaptopurine,Methotrexate; Drug: Methotrexate, 6-mercaptopurine
- Intermediate risk group (Other): Stage III or IV or receiving steroids within one week prior to the diagnosis: Induction protocol I followed by the extracompartmental protocol M, reintensification protocol II, and maintenance therapy for up to a total therapy duration of 104 weeks. Twenty-two triple intrathecal injections.
  Interventions: Drug: Prednisone,Vincristine, Pegylated-asparaginase, Cytarabine, Cyclophosphamide, Daunorubicin, 6-mercaptopurine; Drug: 6-mercaptopurine,Methotrexate; Drug: Dexamethasone,Vincristine, Pegylated-asparaginase, Cytarabine, Cyclophosphamide, Doxorubicin, 6-mercaptopurine; Drug: Methotrexate, 6-mercaptopurine
- High risk group (Other): Failure to qualify a PR, or >5% BM blasts, or with CNS disease on d33 of induction: Induction protocol I followed by 6 intensive polychemotherapy blocks (HR1'-HR2'-HR3'-HR1'-HR2'-HR3'), reintensification protocol II, and maintenance therapy for up to a total therapy duration of 104 weeks. Twenty-two triple intrathecal injections.
  Interventions: Drug: Prednisone,Vincristine, Pegylated-asparaginase, Cytarabine, Cyclophosphamide, Daunorubicin, 6-mercaptopurine; Drug: Dexamethasone,Vincristine, Pegylated-asparaginase, Cytarabine, Cyclophosphamide, Doxorubicin, 6-mercaptopurine; Drug: Dexamethasone,Vincristine, Pegylated-asparaginase, Cytarabine, Cyclophosphamide, Methotrexate; Drug: Dexamethasone, Vindesine, Methotrexate, Ifosfamide, Daunorubicin, Pegylated-asparaginase; Drug: Dexamethasone, Cytarabine, Etoposide, Pegylated-asparaginase; Drug: Methotrexate, 6-mercaptopurine

INTERVENTIONS:
Drug: Prednisone,Vincristine, Pegylated-asparaginase, Cytarabine, Cyclophosphamide, Daunorubicin, 6-mercaptopurine — Prednisone 60 mg/m2 per day,d1-28, then taper over 9 days; Vincristine 1.5 mg/m2 per day (max 2 mg),d1,8, 15, 22; Daunorubicin 30 mg/m2 per dose,d5,12,19; Pegylated-asparaginase 2000 IU/m2 per dose,d16,36,57; Cyclophosphamide 1000 mg/m2 per dose, d36, 57; Cytarabine 75 mg/m2 /d, d36-42,d 57-63; 6-Mercaptopurine 60 mg/m2 per day, d36-42, 57-63; Triple it, d8,29,36,57 1,8, 15, 22
  Other Names: Induction I
Drug: 6-mercaptopurine,Methotrexate — 6-Mercaptopurine 25 mg/m2 per day, d1-56; Methotrexate 5g/m2 per dose, d1, 15, 29, 43; Triple it, d1, 15, 29, 43;
  Other Names: Protocol M
  Arms: Intermediate risk group; Low risk group
Drug: Dexamethasone,Vincristine, Pegylated-asparaginase, Cytarabine, Cyclophosphamide, Doxorubicin, 6-mercaptopurine — Dexamethasone 10 mg/m2 per day, d1-7, d15-21; Vincristine 1.5 mg/m2 per day (max 2 mg), d1, 8, 15; Doxorubicin 30 mg/m2 per dose, d1, 8, 15; Pegylated-asparaginase 2,000 IU/m2 per dose, d3, 24; Cyclophosphamide 1000 mg/m2 per dose, d29; Cytarabine 75 mg/m2 /d, d29-35; 6-Mercaptopurine 60 mg/m2 per day, d29-35; Triple it, d1, 29;
  Other Names: Reinduction II
  Arms: High risk group; Intermediate risk group
Drug: Dexamethasone,Vincristine, Pegylated-asparaginase, Cytarabine, Cyclophosphamide, Methotrexate — Dexamethasone 20mg/m2/day, d1-5; Vincristine 1.5 mg/m2 per day (max 2 mg), d1, 6; Methotrexate 5000mg/m2, d1; Cyclophosphamide 200mg/m2/dose, q12h×5, d2-4; Cytarabine 2000mg/m2/dose, ，q12h×2, d5; Pegylated-asparaginase 2,000 IU/m2 per dose, d6; Triple it, d1;
  Other Names: HR 1'
  Arms: High risk group
Drug: Dexamethasone, Vindesine, Methotrexate, Ifosfamide, Daunorubicin, Pegylated-asparaginase — Dexamethasone 20mg/m2/day, d1-5; Vindesine 3mg/m2（MAX 5mg）, d1, 6; Methotrexate 5000mg/m2, d1; Ifosfamide 800mg/m2/dose, q12h×5,d2-4; Daunorubicin 25mg/m2/dose, d5; Pegylated-asparaginase 2,000 IU/m2 per dose, d6; Triple it, d1;
  Other Names: HR 2'
  Arms: High risk group
Drug: Dexamethasone, Cytarabine, Etoposide, Pegylated-asparaginase — Dexamethasone 20mg/m2/day, d1-5; Cytarabine 2000mg/m2/dose，q12h× 4, d1, 2; Etoposide 100mg/m2/dose，q12h×5, d3,4,5; Pegylated-asparaginase 2,000 IU/m2 per dose, d6; Triple it, d5;
  Other Names: HR 3'
  Arms: High risk group
Drug: Methotrexate, 6-mercaptopurine — 6-mercaptopurine 50 mg/m2 per day, Daily; Methotrexate 20 mg/m2 per dose, Once a week; Triple it, Once every 4 weeks for 12 times;
  Other Names: maintenance therapy

SUMMARY:
The outcomes of children with lymphoblastic lymphoma (LBL) in China in the investigators' previous study were not unexpected. In this study, through further modification treatment protocols and strengthen domestic multicenter collaboration, the investigators try to improve survival for children with LBL when compared to the previous study.

DETAILED DESCRIPTION:
The treatment for LBL is an ALL (acute lymphoblastic leukemia)-based treatment. Additional, high dose L-asparaginase was reported to improve disease-free survival for patients with ALL. The event free survival (EFS) for pediatric LBL in most western countries have achieved 75% to 85%. However, the outcomes of children with LBL in China were not unexpected. In the previous study (CCCG-LBL-2010, 2009-2013), 96 patients with newly diagnosed LBL from 7 Chinese pediatric oncology centers were included. At a median follow-up of 21 months (range, 0.3~60.7months), the 2-year event free survival was 68±5% in all patients. Patients who had achieved complete remission on day 33 of induction had significantly better EFS than those who had not (77±6% v.s.17±10%, p<0.005). In the current trial, the investigators try to improve survival for children with LBL in China through further modification treatment protocols and strengthen domestic multicenter collaboration.

The BFM backbone will be used as the standard backbone therapy for this study. Three doses of daunorubicin are prescribed in induction compared with 4 doses in BFM studies. Cranial radiotherapy only saved for patients (>2 yrs) with CNS disease at presentation.

Complete remission (CR) is defined as at least 75% tumor regression, less than 5% BM (bone marrow)blasts, no CNS (central nervous system) disease, and disappearances of all evidence of disease from all sites for at least 4 weeks. Partial response (PR) is defined as > 50% tumor regression, and no new lesions.Response to treatment is evaluated on day 33 and day 64 of induction.Patients will be stratified into 3 risk groups.

Low risk group: patients (stage I or II) receive induction protocol I followed by the extracompartmental protocol M, and maintenance for up to a total therapy duration of 96 weeks. Totally, 3 doses of PEG-asparaginase (Pegylated-asparaginase) are applied in this group.

Intermediate risk group: patients (stage III or IV or receiving steroids within one week prior to the diagnosis) receive induction protocol I followed by the extracompartmental protocol M, reintensification protocol II, and maintenance for up to a total therapy duration of 104 weeks.Totally, 5 doses of PEG-asparaginase are applied in this group.

High risk group:patients (failure to qualify a PR, or >5% BM blasts, or with CNS disease on d33 of induction) receive induction protocol I followed by 6 intensive polychemotherapy blocks (R'), reintensification protocol II, and maintenance for up to a total therapy duration of 104 weeks. Totally, 11 doses of PEG-asparaginase are applied in this group.

Second look biopsy/resection is indicated for patients without CR on day 64 of induction. Allo- or auto-hematopoietic stem-cell transplantation is recommended for patients with residual tumor. Patients who have disease progression at any time will be removed from this protocol therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed lymphoblastic lymphoma; Patients shall have had no prior cytotoxic chemotherapy with the exception of steroids (<420mg/m2)

Exclusion Criteria:

* Patients with Down syndrome;
* Morphologically unclassifiable lymphoma
* Patients with congenital immunodeficiency, chromosomal breakage syndrome, prior organ transplantation, previous malignancy of any type, or known positive HIV serology.
* Evidence of pregnancy or lactation period.
* Ph+ lymphoblastic lymphoma

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Event free survival for the whole cohort | 3 years
Event free survival for patients in High risk group | 3 years

SECONDARY OUTCOMES:
Overall survival for all patients | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jin Gao, M.D., Principal Investigator — Shanghai Children's Medical Center
Locations (2):
- China (2):
  - West China Second University Hospital, Chengdu
  - Shanghai Children's Medical Center, Shanghai

REFERENCES:
- [Result] Burkhardt B, Reiter A, Landmann E, Lang P, Lassay L, Dickerhoff R, Lakomek M, Henze G, von Stackelberg A. Poor outcome for children and adolescents with progressive disease or relapse of lymphoblastic lymphoma: a report from the berlin-frankfurt-muenster group. J Clin Oncol. 2009 Jul 10;27(20):3363-9. doi: 10.1200/JCO.2008.19.3367. Epub 2009 May 11. PMID 19433688
- [Result] Reiter A, Schrappe M, Ludwig WD, Tiemann M, Parwaresch R, Zimmermann M, Schirg E, Henze G, Schellong G, Gadner H, Riehm H. Intensive ALL-type therapy without local radiotherapy provides a 90% event-free survival for children with T-cell lymphoblastic lymphoma: a BFM group report. Blood. 2000 Jan 15;95(2):416-21. PMID 10627444
- [Result] Moghrabi A, Levy DE, Asselin B, Barr R, Clavell L, Hurwitz C, Samson Y, Schorin M, Dalton VK, Lipshultz SE, Neuberg DS, Gelber RD, Cohen HJ, Sallan SE, Silverman LB. Results of the Dana-Farber Cancer Institute ALL Consortium Protocol 95-01 for children with acute lymphoblastic leukemia. Blood. 2007 Feb 1;109(3):896-904. doi: 10.1182/blood-2006-06-027714. Epub 2006 Sep 26. PMID 17003366
- [Result] Stary J, Zimmermann M, Campbell M, Castillo L, Dibar E, Donska S, Gonzalez A, Izraeli S, Janic D, Jazbec J, Konja J, Kaiserova E, Kowalczyk J, Kovacs G, Li CK, Magyarosy E, Popa A, Stark B, Jabali Y, Trka J, Hrusak O, Riehm H, Masera G, Schrappe M. Intensive chemotherapy for childhood acute lymphoblastic leukemia: results of the randomized intercontinental trial ALL IC-BFM 2002. J Clin Oncol. 2014 Jan 20;32(3):174-84. doi: 10.1200/JCO.2013.48.6522. Epub 2013 Dec 16. PMID 24344215
- [Result] Lymphoma Study Group, Subspecialty Group of Hematology, the Society of Pediatrics, Chinese Medical Association; Lymphoma Study Group Committee of Pediatrics Chinese Anti-Cancer Association. [A collaborative study of children with lymphoblastic non-Hodgkin's lymphoma in China]. Zhonghua Er Ke Za Zhi. 2015 Dec;53(12):931-7. Chinese. PMID 26887549
- [Result] Burkhardt B, Woessmann W, Zimmermann M, Kontny U, Vormoor J, Doerffel W, Mann G, Henze G, Niggli F, Ludwig WD, Janssen D, Riehm H, Schrappe M, Reiter A. Impact of cranial radiotherapy on central nervous system prophylaxis in children and adolescents with central nervous system-negative stage III or IV lymphoblastic lymphoma. J Clin Oncol. 2006 Jan 20;24(3):491-9. doi: 10.1200/JCO.2005.02.2707. PMID 16421426
- [Result] Widjajanto PH, Sumadiono S, Purwanto I, Sutaryo S, Veerman AJ. L-asparaginase: long-term results of a randomized trial of the effect of additional 3 doses during consolidation treatment in the Indonesian WK-ALL-2000 protocol. J Pediatr Hematol Oncol. 2013 Nov;35(8):597-602. doi: 10.1097/MPH.0b013e31827e7f89. PMID 23389497
- [Derived] Yu Q, Wang G, Wang J, Zhang W, Meng L, Cao Y. Primary Testicular and Cutaneous Philadelphia Chromosome Positive B-Cell Lymphoblastic Lymphoma: A Rare Case and Review. Cancer Manag Res. 2022 Apr 21;14:1507-1514. doi: 10.2147/CMAR.S353022. eCollection 2022. PMID 35478711

DOCUMENTS (2):
  • Study Protocol (2017-12-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT02845882/Prot_001.pdf
  • Statistical Analysis Plan (2017-12-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT02845882/SAP_000.pdf